CLINICAL TRIAL: NCT04978402
Title: Management of Insertional Translocation Carriers for Preimplantation Genetic Testing and the Relevance of Sperm Analysis for Reproductive Risk Estimation.
Brief Title: Interchromosomal Insertion Carriers PGT-SR
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0486
Record Dates: First submitted 2021-07-19; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Interchromosomal Breakpoint; Infertility
Keywords: Patients carriers of Insertional translocation (IT); Several years of miscarriages; Abrotions and primary infertility; Interchromosomal insertion; PGT-SR; Sperm.
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Interchromosomal insertions (IT) are rare and complex structural rearrangements. Theoretically, the risk to have a child to term with a malformation or mental retardation can reach 50% related to the proportion of unbalanced gametes produced from behavior of chromosomes during meiosis. However, the meiotic segregation of IT has rarely been studied. This study provide an accurate reproductive risk of IT carriers resulting from a combined analysis of Sperm-FISH and preimplantation genetic testing for structural rearrangement (PGT-SR) management of IT carriers.

ELIGIBILITY:
Inclusion criteria:

- Adult patient whom carrying Insertional translocation in the context of PGT-SR management

Exclusion Criteria:

- Patient who reject the study protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Interchromosomal insertions (IT) are rare and complex structural rearrangements. Theoretically, the risk to have a child to term with a malformation or mental retardation can reach 50% related to the proportion of unbalanced gametes produced from behavior of chromosomes during meiosis.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
estimate the IT carrier's reproductive risk | day 1
  estimate the IT carrier's reproductive risk by investigation of the meiotic segregation of sperm from IT carriers by FISH and evaluate PGT-SR results of male and female IT carriers

CONTACTS AND LOCATIONS:
Overall Officials: Izabel Bernicot, Ph.D, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC